CLINICAL TRIAL: NCT02792699
Title: A Randomized, Double-blind Study to Compare Pharmacokinetics and Pharmacodynamics, Efficacy and Safety of ABP 798 With Rituximab in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: Study to Assess if ABP 798 is Safe & Effective in Treating Moderate to Severe Rheumatoid Arthritis (RA) Compared to Rituximab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20130108; 2013-005543-90 (EudraCT Number)
Record Dates: First submitted 2016-04-25; First posted 2016-06-07 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ABP 798 / ABP 798 (Experimental): Participants received ABP 798 on days 1 and 15 (dose 1) and a second dose of ABP 798 at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
  Interventions: Drug: ABP 798
- Rituximab (US) / ABP 798 (Active Comparator): Participants received rituximab (United States [US] formulation) on days 1 and 15 (dose 1) and transitioned to receive ABP 798 at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
  Interventions: Drug: ABP 798; Drug: Rituximab (US)
- Rituximab (EU) / Rituximab (EU) (Active Comparator): Participants received rituximab (European Union [EU] formulation) on days 1 and 15 (dose 1) and a second dose of rituximab (EU formulation) at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
  Interventions: Drug: Rituximab (EU)

INTERVENTIONS:
Drug: ABP 798 — Supplied as a 10 mg/mL liquid concentrate for intravenous (IV) administration.
  Arms: ABP 798 / ABP 798; Rituximab (US) / ABP 798
Drug: Rituximab (US) — Supplied as a 10 mg/mL liquid concentrate for IV administration.
  Other Names: Rituxan®
  Arms: Rituximab (US) / ABP 798
Drug: Rituximab (EU) — Supplied as a 10 mg/mL liquid concentrate for IV administration.
  Other Names: MabThera®
  Arms: Rituximab (EU) / Rituximab (EU)

SUMMARY:
This trial is designed to determine what effects the human body has on the investigational medicine, ABP 798, and what effects the body has on the investigational medicine after you have been given it, and if this is comparable to what is seen for the licensed medicine, rituximab, in patients with moderate or severe RA.

This study will also assess if the investigational medicine is safe and effective in treating moderate or severe RA compared to the licensed medicine.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 18 and ≤ 80 years old
* Subjects must be diagnosed with rheumatoid arthritis for at least 6 months before baseline
* Active RA defined as ≥ 6 swollen joints and ≥ 6 tender joints at screening and baseline and at least one of the following at screening:

  * erythrocyte sedimentation rate (ESR) ≥ 28 mm/hr
  * serum C-reactive protein (CRP) > 1.0 mg/dL
* Subjects must be taking methotrexate (MTX) for ≥ 12 consecutive weeks and on a stable dose of MTX 7.5 to 25 mg/week for ≥ 8 weeks prior to receiving the investigational product (IP), and be willing to remain on a stable dose throughout the study
* Subject has no known history of active tuberculosis

Exclusion Criteria:

* Class IV RA, Felty's syndrome or history of prosthetic or native joint infection
* Major chronic inflammatory disease or connective tissue disease other than RA, with the exception of secondary Sjögren's syndrome
* Use of commercially available or investigational biologic therapies for RA as follows:

  * anakinra, etanercept within 1 month prior to first dose of IP
  * infliximab, abatacept, tocilizumab, golimumab, certolizumab within 3 months prior to first dose of IP
  * other experimental or commercially available biologic therapies for RA within 3 months or 5 half-lives (whichever is longer) prior to first dose of IP
* Previous receipt of rituximab or a biosimilar of rituximab

Other Inclusion/Exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2016-05-17 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (51):
- United States (27):
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Thousand Oaks, California
  - Research Site, Upland, California
  - Research Site, Aventura, Florida
  - Research Site, Edgewater, Florida
  - Research Site, Hialeah, Florida
  - Research Site, Orlando, Florida
  - Research Site, Vero Beach, Florida
  - Research Site, Idaho Falls, Idaho
  - Research Site, Lexington, Kentucky
  - Research Site, Lansing, Michigan
  - Research Site, Flowood, Mississippi
  - Research Site, Las Vegas, Nevada
  - Research Site, Charlotte, North Carolina
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Duncansville, Pennsylvania
  - Research Site, Orangeburg, South Carolina
  - Research Site, Summerville, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Carrollton, Texas
  - Research Site, Dallas, Texas
  - Research Site, League City, Texas
  - Research Site, Mesquite, Texas
  - Research Site, Plano, Texas
  - Research Site, Olympia, Washington
  - Research Site, Spokane, Washington
- Bulgaria (2):
  - Research Site, Sofia, Sofia
  - Research Site, Plovdiv
- Estonia (2):
  - Research Site, Tallinn, Harjuma
  - Research Site, Tartu
- Germany (3):
  - Research Site, Bad Nauheim, Hesse
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Berlin
- Hungary (5):
  - Research Site, Gyula, Bekes County
  - Research Site, Szentes, Csongrád megye
  - Research Site, Budapest, Pest County
  - Research Site, Szombathely, Vas County
  - Research Site, Veszprém, Veszprém megye
- Poland (12):
  - Research Site, Poznan, Greater Poland Voivodeship
  - Research Site, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Research Site, Krakow, Lesser Poland Voivodeship
  - Research Site, Wroclaw, Lower Silesian Voivodeship
  - Research Site, Lublin, Lublin Voivodeship
  - Research Site, Warsaw, Masovian Voivodeship
  - Research Site, Stalowa Wola, Podkarpackie Voivodeship
  - Research Site, Bialystok, Podlaskie Voivodeship
  - Research Site, Gdansk, Pomeranian Voivodeship
  - Research Site, Katowice, Silesian Voivodeship
  - Research Site, Elblag, Warmian-Masurian Voivodeship
  - Research Site, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Derived] Burmester G, Chien D, Chow V, Gessner M, Pan J, Cohen S. A Randomized, Double-Blind Study Comparing Pharmacokinetics and Pharmacodynamics of Proposed Biosimilar ABP 798 With Rituximab Reference Product in Subjects With Moderate to Severe Rheumatoid Arthritis. Clin Pharmacol Drug Dev. 2020 Nov;9(8):1003-1014. doi: 10.1002/cpdd.845. Epub 2020 Jul 5. PMID 32627420
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 57 centers in Bulgaria, Estonia, Germany, Hungary, Poland, and the United States (US).
  Eligible participants were men and women aged 18 to 80 years, inclusive, with a diagnosis of rheumatoid arthritis (RA) for at least 6 months.
Pre-assignment Details: Participants were randomized in a 1:1:1 ratio to 1 of 3 groups, stratified by geographic region (North America vs Eastern Europe vs Western Europe), seropositivity (rheumatoid factor [RF]-positive and/or cyclic citrullinated peptide [CCP]-positive vs RF-negative and CCP-negative), and number of prior biologic therapies used for RA (1 vs > 1).
Groups:
- Rituximab (EU) / Rituximab (EU): Participants received rituximab (EU formulation) on days 1 and 15 (dose 1) and a second dose of rituximab (EU formulation) at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
- Rituximab (US) / ABP 798: Participants received rituximab (US formulation) on days 1 and 15 (dose 1) and transitioned to receive ABP 798 at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
Period: Overall Study
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Started | 104 | 104 | 103
Received First Infusion of First Dose (Day 1) | 104 | 104 | 103
Received Second Infusion of First Dose (Day 15 (week 2)) | 102 | 103 | 99
Received First Infusion of Second Dose (Week 24) | 97 | 99 | 95
Received Second Infusion of Second Dose (Week 26) | 97 | 99 | 93
Completed | 95 | 94 | 93
Not Completed | 9 | 10 | 10
Not completed — Adverse Event | 1 | 2 | 4
Not completed — Withdrawal by Subject | 4 | 4 | 3
Not completed — Lost to Follow-up | 0 | 1 | 2
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Dissatisfaction with Treatment Efficacy | 1 | 3 | 1
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798 | Total
Number analyzed (Participants) | 104 | 104 | 103 | 311
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.70) | 56.8 (11.34) | 56.4 (10.66) | 55.9 (10.91)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 87 | 74 | 78 | 239
  ≥ 65 years | 17 | 30 | 25 | 72
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 91 | 83 | 264
  Male | 14 | 13 | 20 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 10 | 11 | 29
  Not Hispanic or Latino | 96 | 94 | 92 | 282
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 97 | 99 | 91 | 287
  Black or African American | 5 | 3 | 10 | 18
  Asian | 0 | 2 | 1 | 3
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  Other | 0 | 0 | 1 | 1
Geographic Region [Count of Participants; unit: Participants]
  North America | 38 | 40 | 39 | 117
  Eastern Europe | 59 | 58 | 59 | 176
  Western Europe | 7 | 6 | 5 | 18
Duration of RA [Mean (Standard Deviation); unit: years] | 11.37 (7.400) | 11.69 (7.945) | 12.48 (9.186) | 11.84 (8.194)
Disease Activity Score 28 - C-Reactive Protein (DAS28[CRP]) [Mean (Standard Deviation); unit: scores on a scale] — DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count
  * C-reactive protein (CRP)
  * Patient's global health assessment measured on a 100 mm visual analog scale. DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission. Population: Full analysis set with available data
  scores on a scale
    number analyzed (Participants) | 103 | 102 | 103 | 308
    (all) | 6.09 (1.035) | 5.84 (1.006) | 6.03 (0.997) | 5.99 (1.015)
Seropositivity [Count of Participants; unit: Participants] — Seropositivity defined as rheumatoid factor [RF]-positive and/or cyclic citrullinated peptide [CCP]-positive vs RF-negative and CCP-negative).
  Participants
    RF positive and/or CCP positive | 86 | 88 | 89 | 263
    RF negative and CCP negative | 18 | 16 | 14 | 48
Prior Biologic Use for RA [Count of Participants; unit: Participants]
  One | 62 | 61 | 63 | 186
  More than one | 42 | 43 | 40 | 125

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Serum Concentration-time Curve From Time 0 to Infinity (AUCinf) After the Second Infusion of the First Dose
Description: Area under the serum concentration-time curve from time 0 extrapolated to infinity (AUCinf) following the second infusion of the first dose (day 15). Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method. AUCinf was estimated using the linear trapezoidal rule.
Time Frame: Day 15, pre-dose, end of infusion, and 3, 6, 24, and 48 hours, and 2, 6, and 10 weeks postdose.
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available AUCinf data. Participants with unreliable terminal elimination rate constant values were excluded.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Groups:
- ABP 798: Participants received 1000 mg ABP 798 by intravenous infusion on days 1 and 15 (dose 1).
- Rituximab (EU): Participants received 1000 mg rituximab (EU formulation) by intravenous infusion on days 1 and 15 (dose 1).
- Rituximab (US): Participants received 1000 mg rituximab (US formulation) by intravenous infusion on days 1 and 15 (dose 1).
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 94 | 96 | 94
h*µg/mL | 149398 (36.2) | 172463 (32.9) | 158529 (34.9)
Statistical Analysis 1: Comparison: ABP 798; Test type: Other; Geometric LS Mean = 152371.4 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 2: Comparison: Rituximab (US); Test type: Other; LS Geometric Mean = 159236.0 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 3: Comparison: Rituximab (EU); Test type: Other; LS Geometric Mean = 172213.2 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 4: Comparison: ABP 798 vs Rituximab (US); The geometric mean ratio (GMR) and confidence interval (CI) was estimated from an analysis of covariance (ANCOVA) model adjusted for weight and geographic region. The GMR was obtained by exponentiating the difference of the means on the natural log scale. The CI was obtained by exponentiating the CI for the difference between the means on the log scale; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [US]) for AUCinf was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9569, 90% CI 2-sided [0.8870 to 1.0323]
Statistical Analysis 5: Comparison: ABP 798 vs Rituximab (EU); [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [EU]) for AUCinf was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.8848, 90% CI 2-sided [0.8204 to 0.9542]
Statistical Analysis 6: Comparison: Rituximab (EU) vs Rituximab (US); [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — PK similarity between the test (rituximab [US]) and reference (rituximab [EU]) for AUCinf was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9246, 90% CI 2-sided [0.8575 to 0.9970]

2. Primary Outcome: Maximum Observed Drug Concentration (Cmax) After the Second Infusion of the First Dose
Description: Maximum observed concentration following the second infusion of the first dose (day 15). Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: Day 15, pre-dose, end of infusion, and 3, 6, 24, and 48 hours, and 2, 6, and 10 weeks postdose.
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available Cmax data on day 15.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 96 | 97 | 93
µg/mL | 361 (23.5) | 394 (22.0) | 372 (24.7)
Statistical Analysis 1: Comparison: ABP 798; Test type: Other; Geometric LS Mean = 368.43 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 2: Comparison: Rituximab (US); Test type: Other; LS Geometric Mean = 374.44 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 3: Comparison: Rituximab (EU); Test type: Other; LS Geometric Mean = 393.29 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 4: Comparison: ABP 798 vs Rituximab (US); [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [US]) for Cmax was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9840, 90% CI 2-sided [0.9356 to 1.0348]
Statistical Analysis 5: Comparison: ABP 798 vs Rituximab (EU); [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [EU]) for Cmax was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9368, 90% CI 2-sided [0.8912 to 0.9848]
Statistical Analysis 6: Comparison: Rituximab (EU) vs Rituximab (US); [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — PK similarity between the test (rituximab [US]) and reference (rituximab [EU]) for Cmax was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9521, 90% CI 2-sided [0.9055 to 1.0010]

3. Secondary Outcome: Area Under the Serum Concentration-time Curve From Predose on Day 1 to 14 Days Postdose (AUC0-14day)
Description: Area under the serum concentration-time curve from time 0 on day 1 prior to the first infusion of the first dose to 14 days postdose. Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method. AUC0-14day was estimated using the linear trapezoidal rule.
Time Frame: Day 1, predose, at end of infusion, 3, 6, 24, and 48 hours postdose and day 15, predose.
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available AUC0-14day data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 98 | 97 | 93
h*µg/mL | 41445 (28.8) | 45161 (24.7) | 43291 (29.6)
Statistical Analysis 1: Comparison: ABP 798; Test type: Other; Geometric LS Mean = 42203.8 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 2: Comparison: Rituximab (US); Test type: Other; LS Geometric Mean = 43378.8 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 3: Comparison: Rituximab (EU); Test type: Other; LS Geometric Mean = 44925.3 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 4: Comparison: ABP 798 vs Rituximab (US); [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [US]) for AUC0-14day was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9729, 90% CI 2-sided [0.9174 to 1.0318]
Statistical Analysis 5: Comparison: ABP 798 vs Rituximab (EU); The geometric mean ratio (GMR) and confidence interval (CI) was estimated from an analysis of covariance ANCOVA model adjusted for weight and geographic region. The GMR was obtained by exponentiating the difference of the means on the natural log scale. The CI was obtained by exponentiating the CI for the difference between the means on the log scale; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [EU]) for AUC0-14day was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9394, 90% CI 2-sided [0.8863 to 0.9958]
Statistical Analysis 6: Comparison: Rituximab (EU) vs Rituximab (US); The geometric mean ratio (GMR) and confidence interval (CI) was estimated from an ANCOVA model adjusted for weight and geographic region. The GMR was obtained by exponentiating the difference of the means on the natural log scale. The CI was obtained by exponentiating the CI for the difference between the means on the log scale; Test type: Equivalence — PK similarity between the test (rituximab [US]) and reference (rituximab [EU]) for AUC0-14day was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9656, 90% CI 2-sided [0.9104 to 1.0240]

4. Secondary Outcome: Area Under the Serum Concentration-time Curve From Predose on Day 1 to Week 12 (AUC0-12wk)
Description: Area under the serum concentration-time curve from time 0 on day 1 prior to the first infusion of the first dose to week 12. Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method. AUC0-12wk was estimated using the linear trapezoidal rule.
Time Frame: Day 1, predose, at end of infusion, 3, 6, 24, and 48 hours postdose; day 15, predose, end of infusion, 3, 6, 24, and 48 hour postdose, and at days 29, 57, and 85 (week 12).
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available AUC0-12wk data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*µg/mL
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 99 | 100 | 96
h*µg/mL | 146369 (34.3) | 166995 (30.5) | 155240 (33.7)
Statistical Analysis 1: Comparison: ABP 798; Test type: Other; Geometric LS Mean = 149590.5 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 2: Comparison: Rituximab (US); Test type: Other; LS Geometric Mean = 155778.7 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 3: Comparison: Rituximab (EU); Test type: Other; LS Geometric Mean = 166811.0 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 4: Comparison: ABP 798 vs Rituximab (US); [analysis description as in outcome 1, analysis 4]; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [US]) for AUC0-12wk was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9603, 90% CI 2-sided [0.8950 to 1.0303]
Statistical Analysis 5: Comparison: ABP 798 vs Rituximab (EU); [analysis description as in outcome 3, analysis 5]; Test type: Equivalence — PK similarity between the test (ABP 798) and reference (rituximab [EU]) for AUC0-12wk was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.8968, 90% CI 2-sided [0.8363 to 0.9616]
Statistical Analysis 6: Comparison: Rituximab (EU) vs Rituximab (US); [analysis description as in outcome 3, analysis 6]; Test type: Equivalence — PK similarity between the test (rituximab [US]) and reference (rituximab [EU]) for AUC0-12wk was demonstrated if the 90% CI for the GMR following the second infusion of the first dose was within the bioequivalence criteria of 0.8 to 1.25; Geometric Mean Ratio = 0.9339, 90% CI 2-sided [0.8707 to 1.0016]

5. Secondary Outcome: Maximum Observed Drug Concentration (Cmax) After the First Infusion of the First Dose
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: Day 1, predose, at end of infusion, 3, 6, 24, and 48 hours postdose and day 15, predose.
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 103 | 103 | 99
µg/mL | 298 (26.1) | 321 (21.2) | 304 (25.5)
Statistical Analysis 1: Comparison: ABP 798; Test type: Other; Geometric LS Mean = 304.04 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 2: Comparison: Rituximab (US); Test type: Other; LS Geometric Mean = 305.80 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 3: Comparison: Rituximab (EU); Test type: Other; LS Geometric Mean = 320.87 — Estimated using an analysis of covariance model adjusted for weight and geographic region
Statistical Analysis 4: Comparison: ABP 798 vs Rituximab (US); [analysis description as in outcome 3, analysis 6]; Test type: Equivalence — [test comment as in outcome 2, analysis 4]; Geometric Mean Ratio = 0.9942, 90% CI 2-sided [0.9461 to 1.0448]
Statistical Analysis 5: Comparison: ABP 798 vs Rituximab (EU); [analysis description as in outcome 3, analysis 6]; Test type: Equivalence — [test comment as in outcome 2, analysis 5]; Geometric Mean Ratio = 0.9475, 90% CI 2-sided [0.9021 to 0.9953]
Statistical Analysis 6: Comparison: Rituximab (EU) vs Rituximab (US); [analysis description as in outcome 3, analysis 6]; Test type: Equivalence — [test comment as in outcome 2, analysis 6]; Geometric Mean Ratio = 0.9531, 90% CI 2-sided [0.9070 to 1.0015]

6. Secondary Outcome: Time of Maximum Observed Drug Concentration (Tmax) After the First and Second Infusions of the First Dose
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: Day 1, predose, at end of infusion, 3, 6, 24, and 48 hours postdose; day 15, predose, end of infusion, 3, 6, 24, and 48 hours postdose, and at days 29, 57, and 85 (week 12).
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available Tmax data at each time point.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 103 | 103 | 99
hours
  After First Infusion (Day 1) | 4.50 [4.35 to 7.18] | 4.67 [4.38 to 7.30] | 4.68 [4.38 to 7.50]
  After Second Infusion (Day 15): number analyzed (Participants) | 96 | 97 | 93
  After Second Infusion (Day 15) | 3.57 [3.42 to 6.03] | 3.67 [3.40 to 5.50] | 4.12 [3.42 to 6.55]

7. Secondary Outcome: Last Measurable Serum Concentration After the Second Infusion up to Week 12 (Clast)
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: Day 15, predose, end of infusion, 3, 6, 24, and 48 hours postdose, and at days 29, 57, and 85 (week 12).
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available Clast data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 101 | 103 | 98
µg/mL | 5.95 (154) | 8.52 (145) | 6.76 (143)

8. Secondary Outcome: Terminal Elimination Half-life (t1/2)
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: as for outcome 6
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available T1/2 data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 96 | 98 | 96
hours | 335.62 (38) | 375.26 (32) | 334.57 (40)

9. Secondary Outcome: Terminal Elimination Rate Constant (λz)
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: Day 1, predose, at end of infusion, 3, 6, 24, and 48 hours postdose; day 15, predose, end of infusion, 3, 6, 24, and 48 hours postdose, and at days 29, 57 and 85 (week 12).
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available λz data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 101 | 103 | 98
1/h | 0.00205 (38.61018) | 0.00187 (33.44044) | 0.00205 (40.15779)

10. Secondary Outcome: Clearance (CL)
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: as for outcome 6
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available CL data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 94 | 96 | 94
L/h | 0.01339 (36.22558) | 0.01160 (32.94524) | 0.01262 (34.93316)

11. Secondary Outcome: Mean Residence Time (MRT)
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: as for outcome 6
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available MRT data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 94 | 96 | 94
hours | 549 (26.7) | 592 (26.5) | 557 (26.8)

12. Secondary Outcome: Percent of AUC Extrapolation (AUC%Extrap)
Description: Percent of AUC extrapolated to infinity in AUCinf. Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: Day 15, predose, end of infusion, 3, 6, 24, and 48 hours postdose, and at days 29, 57, and 85 (week 12).
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available AUC%extrap data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent extrapolation
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 101 | 103 | 98
percent extrapolation | 1.91 (161) | 2.62 (146) | 2.06 (148)

13. Secondary Outcome: AUC0-12 wk/AUCinf
Description: Concentrations of ABP-798 and rituximab were quantified using a validated electrochemiluminescent method.
Time Frame: as for outcome 6
Population: The pharmacokinetic (PK) parameter analysis set (randomized participants who received the full protocol-specified infusion on day 1 and had an evaluable ABP 798 or rituximab serum concentration-time profile) with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 96 | 98 | 96
ratio | 0.97 (3) | 0.96 (4) | 0.97 (3)

14. Secondary Outcome: Change From Baseline in Disease Activity Score 28-CRP at Week 24
Description: The DAS28 measures the severity of disease at a specific time and is derived from the following variables:
  * 28 tender joint count
  * 28 swollen joint count
  * C-reactive protein (CRP)
  * Patient's global health assessment measured on a 100 mm VAS, where 0 mm = no RA activity and 100 mm = worst RA activity imaginable.
  DAS28(CRP) scores range from 0 to approximately 10, with the upper bound dependent on the highest possible level of CRP. A DAS28 score higher than 5.1 indicates high disease activity, a DAS28 score less than 3.2 indicates low disease activity, and a DAS28 score less than 2.6 indicates clinical remission.
Time Frame: Baseline and Week 24
Population: Full analysis set with observed data conducted using a repeated measures analysis in which data from all assessed postbaseline time points were included.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Rituximab (US + EU): Participants received 1000 mg rituximab (US or EU formulation) on days 1 and 15 (dose 1) by intravenous infusion.
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US) | Rituximab (US + EU)
Number analyzed (Participants) | 104 | 104 | 103 | 207
units on a scale | -2.006 (0.1313) | -2.116 (0.1339) | -1.936 (0.1349) | -2.026 (0.1039)
Statistical Analysis 1: Comparison: ABP 798 vs Rituximab (US + EU); If PK similarity was established between rituximab (US) and rituximab (EU), the 2 rituximab arms were to be combined into a single reference group for the primary assessment of clinical equivalence of DAS28-CRP change from baseline at week 24 using a repeated measures analysis with DAS28-CRP change from baseline as the response and the stratification variables, visit, treatment, treatment-by-visit interaction and baseline DAS28-CRP as predictors, and unstructured covariance matrix in the model; Test type: Equivalence — Clinical equivalence was tested by comparing the 2-sided 90% CI of the change from baseline at week 24 of DAS28-CRP between ABP 798 and rituximab with an equivalence margin of (-0.6, 0.6); LS Mean Difference = 0.020, 90% CI 2-sided [-0.225 to 0.264]
Statistical Analysis 2: Comparison: ABP 798 vs Rituximab (US); Test type: Other; LS Mean Difference = -0.070, 90% CI 2-sided [-0.353 to 0.213]
Statistical Analysis 3: Comparison: ABP 798 vs Rituximab (EU); Test type: Other; LS Mean Difference = 0.110, 90% CI 2-sided [-0.171 to 0.392]

15. Secondary Outcome: Change From Baseline in Disease Activity Score 28-CRP at Weeks 8, 12, 40, and 48
Description: as for outcome 14
Time Frame: Baseline and weeks 8, 12, 40, and 48
Population: Full analysis set with observed data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 104 | 104 | 103
units on a scale
  Week 8: number analyzed (Participants) | 98 | 94 | 96
  Week 8 | -1.674 (0.1259) | -1.738 (0.1335) | -1.527 (0.1330)
  Week 12: number analyzed (Participants) | 95 | 98 | 95
  Week 12 | -1.746 (0.1302) | -2.248 (0.1357) | -2.016 (0.1367)
  Week 40: number analyzed (Participants) | 93 | 93 | 92
  Week 40 | -2.038 (0.1440) | -2.293 (0.1494) | -2.198 (0.1489)
  Week 48: number analyzed (Participants) | 86 | 83 | 89
  Week 48 | -2.243 (0.1473) | -2.505 (0.1553) | -2.323 (0.1486)
Statistical Analysis 1: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of change from baseline at week 8, based on an ANCOVA model adjusted for baseline DAS28-CRP and the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = 0.064, 90% CI 2-sided [-0.203 to 0.330]
Statistical Analysis 2: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 15, analysis 1]; Test type: Other; LS Mean Difference = -0.147, 90% CI 2-sided [-0.411 to 0.117]
Statistical Analysis 3: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of change from baseline at week 12, based on an ANCOVA model adjusted for baseline DAS28-CRP and the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = 0.502, 90% CI 2-sided [0.233 to 0.772]
Statistical Analysis 4: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 15, analysis 3]; Test type: Other; LS Mean Difference = 0.270, 90% CI 2-sided [0.000 to 0.539]
Statistical Analysis 5: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of change from baseline at week 40, based on an ANCOVA model adjusted for baseline DAS28-CRP and the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = 0.255, 90% CI 2-sided [-0.040 to 0.550]
Statistical Analysis 6: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 15, analysis 5]; Test type: Other; LS Mean Difference = 0.160, 90% CI 2-sided [-0.135 to 0.455]
Statistical Analysis 7: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of change from baseline at week 48, based on an ANCOVA model adjusted for baseline DAS28-CRP and the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = 0.262, 90% CI 2-sided [-0.040 to 0.564]
Statistical Analysis 8: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 15, analysis 7]; Test type: Other; LS Mean Difference = 0.080, 90% CI 2-sided [-0.216 to 0.376]

16. Secondary Outcome: Percentage of Participants With an ACR20 Response
Description: A positive ACR20 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 20% improvement in 68 tender joint count;
  * ≥ 20% improvement in 66 swollen joint count; and
  * ≥ 20% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of disease-related pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global health assessment (measured on a 100 mm VAS);
    * Investigator's global health assessment (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and Weeks 8, 12, 24, 40, and 48
Population: Full analysis set with observed data
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 104 | 104 | 103
percentage of participants
  Week 8: number analyzed (Participants) | 101 | 100 | 97
  Week 8 | 56.4 | 60.0 | 54.6
  Week 12: number analyzed (Participants) | 102 | 101 | 98
  Week 12 | 67.6 | 73.3 | 63.3
  Week 24: number analyzed (Participants) | 99 | 102 | 95
  Week 24 | 70.7 | 66.7 | 64.2
  Week 40: number analyzed (Participants) | 93 | 95 | 91
  Week 40 | 68.8 | 73.7 | 68.1
  Week 48: number analyzed (Participants) | 87 | 84 | 88
  Week 48 | 63.2 | 79.8 | 75.0
Statistical Analysis 1: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk ratio (ABP 798/ABP 798 versus Rituximab [EU]/Rituximab [EU]) at week 8, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 0.9339, 90% CI 2-sided [0.7696 to 1.1332]
Statistical Analysis 2: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 8, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = -0.0360, 90% CI 2-sided [-0.1495 to 0.0775]
Statistical Analysis 3: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk ratio (ABP 798/ABP 798 versus Rituximab [US]/ABP 798]) at week 8, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 1.0392, 90% CI 2-sided [0.8436 to 1.2801]
Statistical Analysis 4: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 8, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = 0.0246, 90% CI 2-sided [-0.0910 to 0.1402]
Statistical Analysis 5: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk ratio (ABP 798/ABP 798 versus Rituximab [EU]/Rituximab [EU]) at week 12, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 0.8780, 90% CI 2-sided [0.7573 to 1.0179]
Statistical Analysis 6: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 12, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = -0.0794, 90% CI 2-sided [-0.1834 to 0.0247]
Statistical Analysis 7: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk ratio (ABP 798/ABP 798 versus Rituximab [US]/ABP 798]) at week 12, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 1.0426, 90% CI 2-sided [0.8770 to 1.2394]
Statistical Analysis 8: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 12, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = 0.0348, 90% CI 2-sided [-0.0758 to 0.1454]
Statistical Analysis 9: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk ratio (ABP 798/ABP 798 versus Rituximab [EU]/Rituximab [EU]) at week 24, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 1.0102, 90% CI 2-sided [0.8743 to 1.1671]
Statistical Analysis 10: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 24, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = 0.0199, 90% CI 2-sided [-0.0835 to 0.1234]
Statistical Analysis 11: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk ratio (ABP 798/ABP 798 versus Rituximab [US]/ABP 798]) at week 24, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 1.0793, 90% CI 2-sided [0.9244 to 1.2601]
Statistical Analysis 12: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 24, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = 0.0561, 90% CI 2-sided [-0.0493 to 0.1615]
Statistical Analysis 13: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk ratio (ABP 798/ABP 798 versus Rituximab [EU]/Rituximab [EU]) at week 40, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 0.8848, 90% CI 2-sided [0.7759 to 1.0091]
Statistical Analysis 14: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 40, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = -0.0776, 90% CI 2-sided [-0.1789 to 0.0237]
Statistical Analysis 15: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk ratio (ABP 798/ABP 798 versus Rituximab [US]/ABP 798]) at week 40, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 0.9982, 90% CI 2-sided [0.8585 to 1.1605]
Statistical Analysis 16: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 40, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = 0.0008, 90% CI 2-sided [-0.1038 to 0.1054]
Statistical Analysis 17: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk ratio (ABP 798/ABP 798 versus Rituximab [EU]/Rituximab [EU]) at week 48, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 0.7862, 90% CI 2-sided [0.6722 to 0.9196]
Statistical Analysis 18: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Risk difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 48, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = -0.2004, 90% CI 2-sided [-0.3066 to -0.0941]
Statistical Analysis 19: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk ratio (ABP 798/ABP 798 versus Rituximab [US]/ABP 798]) at week 48, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Ratio (RR) = 0.8804, 90% CI 2-sided [0.7587 to 1.0215]
Statistical Analysis 20: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Risk difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 48, based on a generalized linear model adjusted for the stratification factors geographic region, seropositivity, and number of prior biologic therapies used for RA as covariates; Test type: Other; Risk Difference (RD) = -0.1037, 90% CI 2-sided [-0.2066 to -0.0007]

17. Secondary Outcome: Percentage of Participants With an ACR50 Response
Description: A positive ACR50 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 50% improvement in 68 tender joint count;
  * ≥ 50% improvement in 66 swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of disease-related pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global health assessment (measured on a 100 mm VAS);
    * Investigator's global health assessment (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and Weeks 8, 12, 24, 40, and 48
Population: Full analysis set with observed data
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 104 | 104 | 103
percentage of participants
  Week 8: number analyzed (Participants) | 101 | 99 | 97
  Week 8 | 26.7 | 29.3 | 24.7
  Week 12: number analyzed (Participants) | 102 | 101 | 98
  Week 12 | 36.3 | 47.5 | 32.7
  Week 24: number analyzed (Participants) | 98 | 102 | 96
  Week 24 | 39.8 | 39.2 | 38.5
  Week 40: number analyzed (Participants) | 94 | 95 | 92
  Week 40 | 48.9 | 57.9 | 45.7
  Week 48: number analyzed (Participants) | 86 | 84 | 88
  Week 48 | 51.2 | 58.3 | 48.9
Statistical Analysis 1: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 1]; Test type: Other; Risk Ratio (RR) = 0.9256, 90% CI 2-sided [0.6400 to 1.3388]
Statistical Analysis 2: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 2]; Test type: Other; Risk Difference (RD) = -0.0181, 90% CI 2-sided [-0.1209 to 0.0847]
Statistical Analysis 3: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 3]; Test type: Other; Risk Ratio (RR) = 1.0868, 90% CI 2-sided [0.7328 to 1.6119]
Statistical Analysis 4: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 4]; Test type: Other; Risk Difference (RD) = 0.0201, 90% CI 2-sided [-0.0803 to 0.1205]
Statistical Analysis 5: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 5]; Test type: Other; Risk Ratio (RR) = 0.7095, 90% CI 2-sided [0.5387 to 0.9346]
Statistical Analysis 6: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 6]; Test type: Other; Risk Difference (RD) = -0.1109, 90% CI 2-sided [-0.2231 to 0.0013]
Statistical Analysis 7: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 7]; Test type: Other; Risk Ratio (RR) = 1.0882, 90% CI 2-sided [0.7829 to 1.5127]
Statistical Analysis 8: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 8]; Test type: Other; Risk Difference (RD) = 0.0441, 90% CI 2-sided [-0.0626 to 0.1508]
Statistical Analysis 9: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 9]; Test type: Other; Risk Ratio (RR) = 0.9612, 90% CI 2-sided [0.7273 to 1.2705]
Statistical Analysis 10: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 10]; Test type: Other; Risk Difference (RD) = 0.0020, 90% CI 2-sided [-0.1081 to 0.1122]
Statistical Analysis 11: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 11]; Test type: Other; Risk Ratio (RR) = 1.0029, 90% CI 2-sided [0.7560 to 1.3305]
Statistical Analysis 12: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 12]; Test type: Other; Risk Difference (RD) = 0.0039, 90% CI 2-sided [-0.1056 to 0.1135]
Statistical Analysis 13: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 13]; Test type: Other; Risk Ratio (RR) = 0.8373, 90% CI 2-sided [0.6797 to 1.0316]
Statistical Analysis 14: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 14]; Test type: Other; Risk Difference (RD) = -0.0863, 90% CI 2-sided [-0.2029 to 0.0302]
Statistical Analysis 15: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 15]; Test type: Other; Risk Ratio (RR) = 1.1191, 90% CI 2-sided [0.8780 to 1.4264]
Statistical Analysis 16: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 16]; Test type: Other; Risk Difference (RD) = 0.0288, 90% CI 2-sided [-0.0827 to 0.1402]
Statistical Analysis 17: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 17]; Test type: Other; Risk Ratio (RR) = 0.8376, 90% CI 2-sided [0.6807 to 1.0307]
Statistical Analysis 18: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 18]; Test type: Other; Risk Difference (RD) = -0.0781, 90% CI 2-sided [-0.2014 to 0.0452]
Statistical Analysis 19: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 19]; Test type: Other; Risk Ratio (RR) = 1.0548, 90% CI 2-sided [0.8351 to 1.3321]
Statistical Analysis 20: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 20]; Test type: Other; Risk Difference (RD) = 0.0141, 90% CI 2-sided [-0.1021 to 0.1303]

18. Secondary Outcome: Percentage of Participants With an ACR70 Response
Description: A positive ACR70 response is defined if the following 3 criteria for improvement from baseline were met:
  * ≥ 70% improvement in 68 tender joint count;
  * ≥ 70% improvement in 66 swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of disease-related pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global health assessment (measured on a 100 mm VAS);
    * Investigator's global health assessment (measured on a 100 mm VAS);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein concentration.
Time Frame: Baseline and Weeks 8, 12, 24, 40, and 48
Population: Full analysis set with observed data
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 104 | 104 | 103
percentage of participants
  Week 8: number analyzed (Participants) | 101 | 100 | 97
  Week 8 | 6.9 | 12.0 | 9.3
  Week 12: number analyzed (Participants) | 101 | 101 | 98
  Week 12 | 12.9 | 19.8 | 16.3
  Week 24: number analyzed (Participants) | 99 | 102 | 96
  Week 24 | 19.2 | 19.6 | 16.7
  Week 40: number analyzed (Participants) | 94 | 94 | 92
  Week 40 | 27.7 | 27.7 | 22.8
  Week 48: number analyzed (Participants) | 87 | 84 | 89
  Week 48 | 28.7 | 39.3 | 24.7
Statistical Analysis 1: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 1]; Test type: Other; Risk Ratio (RR) = 0.5926, 90% CI 2-sided [0.2818 to 1.2462]
Statistical Analysis 2: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 2]; Test type: Other; Risk Difference (RD) = -0.0574, 90% CI 2-sided [-0.1285 to 0.0136]
Statistical Analysis 3: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 3]; Test type: Other; Risk Ratio (RR) = 0.7476, 90% CI 2-sided [0.3383 to 1.6519]
Statistical Analysis 4: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 4]; Test type: Other; Risk Difference (RD) = -0.0327, 90% CI 2-sided [-0.0962 to 0.0308]
Statistical Analysis 5: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 5]; Test type: Other; Risk Ratio (RR) = 0.6346, 90% CI 2-sided [0.3704 to 1.0872]
Statistical Analysis 6: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 6]; Test type: Other; Risk Difference (RD) = -0.0569, 90% CI 2-sided [-0.1448 to 0.0310]
Statistical Analysis 7: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 7]; Test type: Other; Risk Ratio (RR) = 0.7857, 90% CI 2-sided [0.4450 to 1.3874]
Statistical Analysis 8: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 8]; Test type: Other; Risk Difference (RD) = -0.0417, 90% CI 2-sided [-1237 to 0.0403]
Statistical Analysis 9: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 9]; Test type: Other; Risk Ratio (RR) = 0.9254, 90% CI 2-sided [0.5772 to 1.4838]
Statistical Analysis 10: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 10]; Test type: Other; Risk Difference (RD) = 0.0156, 90% CI 2-sided [-0.0780 to 0.1092]
Statistical Analysis 11: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 11]; Test type: Other; Risk Ratio (RR) = 1.1120, 90% CI 2-sided [0.6722 to 1.8398]
Statistical Analysis 12: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 12]; Test type: Other; Risk Difference (RD) = 0.0244, 90% CI 2-sided [-0.0630 to 0.1119]
Statistical Analysis 13: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 13]; Test type: Other; Risk Ratio (RR) = 0.9798, 90% CI 2-sided [0.6675 to 1.4384]
Statistical Analysis 14: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 14]; Test type: Other; Risk Difference (RD) = 0.0375, 90% CI 2-sided [-0.0707 to 0.1456]
Statistical Analysis 15: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 15]; Test type: Other; Risk Ratio (RR) = 1.1831, 90% CI 2-sided [0.7833 to 1.7870]
Statistical Analysis 16: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 16]; Test type: Other; Risk Difference (RD) = 0.0752, 90% CI 2-sided [-0.0297 to 0.1802]
Statistical Analysis 17: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 17]; Test type: Other; Risk Ratio (RR) = 0.7027, 90% CI 2-sided [0.4930 to 1.0017]
Statistical Analysis 18: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); [analysis description as in outcome 16, analysis 18]; Test type: Other; Risk Difference (RD) = -0.0908, 90% CI 2-sided [-0.2110 to 0.0294]
Statistical Analysis 19: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 19]; Test type: Other; Risk Ratio (RR) = 1.1449, 90% CI 2-sided [0.7601 to 1.7246]
Statistical Analysis 20: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; [analysis description as in outcome 16, analysis 20]; Test type: Other; Risk Difference (RD) = 0.0277, 90% CI 2-sided [-0.0804 to 0.1357]

19. Secondary Outcome: Hybrid ACR
Description: The hybrid ACR combines the ACR 20/50/70 response with the mean percent change in all 7 ACR core components, thus providing a percent improvement from baseline on a continuous scale. For each participant, the mean percent improvement from baseline across the 7 ACR core set measures (tender joint count, swollen joint count, Patient's Global Assessment of Disease Activity, Investigator's Global Assessment of Disease Activity, disability index of the HAQ, and CRP) was calculated (a positive change indicates improvement, and the maximum worst change is limited to -100%) and the ACR20, ACR50, and ACR70 response is determined. The hybrid ACR is determined from a reference table taking into account both ACR response and mean percent improvement in the core set measures. Scores can range from -100% (maximal worsening) to 100% (maximal improvement).
Time Frame: Baseline and weeks 8, 12, 24, 40, and 48
Population: Full analysis set with observed data
Measure: Least Squares Mean (Standard Error); unit: percent improvement
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 104 | 104 | 103
percent improvement
  Week 8: number analyzed (Participants) | 94 | 95 | 92
  Week 8 | 32.631 (2.7287) | 34.630 (2.8058) | 32.086 (2.8628)
  Week 12: number analyzed (Participants) | 98 | 101 | 94
  Week 12 | 36.604 (2.8910) | 44.828 (2.9412) | 38.664 (3.0360)
  Week 24: number analyzed (Participants) | 94 | 100 | 93
  Week 24 | 39.269 (3.1660) | 40.589 (3.1781) | 38.539 (3.2436)
  Week 40: number analyzed (Participants) | 91 | 94 | 89
  Week 40 | 41.042 (3.1508) | 43.250 (3.1916) | 41.078 (3.2459)
  Week 48: number analyzed (Participants) | 85 | 84 | 87
  Week 48 | 41.917 (3.3878) | 48.546 (3.4870) | 45.013 (3.3942)
Statistical Analysis 1: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 8, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -1.999, 90% CI 2-sided [-7.673 to 3.675]
Statistical Analysis 2: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 8, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = 0.544, 90% CI 2-sided [-5.185 to 6.274]
Statistical Analysis 3: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 12, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -8.224, 90% CI 2-sided [-14.102 to -2.346]
Statistical Analysis 4: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 12, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -2.060, 90% CI 2-sided [-8.052 to 3.933]
Statistical Analysis 5: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 24, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -1.320, 90% CI 2-sided [-7.620 to 4.979]
Statistical Analysis 6: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 24, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = 0.730, 90% CI 2-sided [-5.691 to 7.150]
Statistical Analysis 7: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 40, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -2.207, 90% CI 2-sided [-8.562 to 1.417]
Statistical Analysis 8: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 40, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -0.036, 90% CI 2-sided [-6.497 to 6.424]
Statistical Analysis 9: Comparison: ABP 798 / ABP 798 vs Rituximab (EU) / Rituximab (EU); Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [EU]/Rituximab [EU]) at week 48, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -6.629, 90% CI 2-sided [-13.455 to 0.197]
Statistical Analysis 10: Comparison: ABP 798 / ABP 798 vs Rituximab (US) / ABP 798; Analysis of the LS mean difference (ABP 798/ABP 798 - Rituximab [US]/ABP 798) at week 48, based on an ANCOVA model adjusted for the stratification variables geographic region, seropositivity, and number of prior biologic therapies used for RA; Test type: Other; LS Mean Difference = -3.096, 90% CI 2-sided [-9.883 to 3.691]

20. Secondary Outcome: Percentage of Participants With Complete Depletion in CD19+ Cell Count on Day 3
Description: Complete depletion of cluster of differentiation (CD) 19 positive cells was defined as a CD19+ cell count < 20 cell/μL (0.02 x 10⁹ cell/L).
Time Frame: Day 3
Population: Full analysis set participants with a day 3 CD19+ cell count; participants with missing CD19+ cell counts at baseline or with CD19+ cell count < 20 cell/μL at baseline were excluded from the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 97 | 96 | 97
percentage of participants | 94.8 | 96.9 | 92.8
Statistical Analysis 1: Comparison: ABP 798 vs Rituximab (EU); Test type: Other; Risk Difference (RD) = -0.0245, 90% CI 2-sided [-0.1083 to 0.0593] — Based on a generalized linear model adjusted for geographic region, seropositivity and prior biologic use as covariates in the model
Statistical Analysis 2: Comparison: ABP 798 vs Rituximab (US); Test type: Other; Risk Difference (RD) = 0.0187, 90% CI 2-sided [-0.0610 to 0.0984] — [estimate comment as in outcome 20, analysis 1]

21. Secondary Outcome: Duration of Complete Depletion in CD19+ Cell Count
Description: Duration of CD19+ B-cell complete depletion was defined as the time from the first incidence of complete depletion of CD19+ cell count (CD19+ cell count < 20 cells/μL) to when the CD19+ cell count first increased to ≥ 20 cells/μL. Participants whose CD19+ cell count did not increase to ≥ 20 cells/μL were censored at the last CD19+ assessment date.
Time Frame: CD19+ cell count was assessed at baseline, days 2, 3, weeks 4, 24, and 48
Population: Full analysis set participants who had a CD19+ complete depletion for at least one postdose time point.
Measure: Median (90% Confidence Interval); unit: days
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 95 | 99 | 98
days | NA [NA to NA] — Could not be estimated due to the low number of events | NA [377.0 to NA] — Could not be estimated due to the low number of events | NA [338.0 to NA] — Could not be estimated due to the low number of events

22. Secondary Outcome: Number of Participants With Adverse Events After the First Dose
Description: Adverse events (AEs) were graded by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 4.03, where Grade 1 = mild AE, Grade 2 = moderate AE, Grade 3 = severe AE, Grade 4 = life-threatening AE, and Grade 5 = death due to AE.
  A serious AE (SAE) was defined as an AE that met at least 1 of the following serious criteria:
  * fatal
  * life-threatening
  * required inpatient hospitalization or prolongation of existing hospitalization
  * resulted in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event. The adverse events of interest prespecified for this study included infusion reactions including hypersensitivity, cardiac disorders, serious infections, progressive multifocal leukoencephalopathy, hematological reactions, hepatitis B reactivation, opportunistic infections, hypogammaglobulinemia, severe mucocutaneous reactions, and gastrointestinal perforation.
Time Frame: From day 1 until the first infusion of the second dose (week 24)
Population: All randomized participants who received at least 1 infusion of study drug (safety analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 798 | Rituximab (EU) | Rituximab (US)
Number analyzed (Participants) | 104 | 104 | 103
Participants
  Any adverse event | 52 | 44 | 44
  Any grade ≥ 3 adverse event | 4 | 6 | 4
  Any fatal adverse event | 0 | 0 | 0
  Any serious adverse event | 4 | 5 | 5
  Any AE leading to discontinuation of drug/study | 3 | 1 | 4
  Any AE leading to infusion delayed/ not given | 6 | 6 | 7
  Any adverse event of interest | 19 | 11 | 18

23. Secondary Outcome: Number of Participants Who Developed Anti-drug Antibodies
Description: Samples were first tested in an electrochemiluminescence (ECL)-based bridging immunoassay to detect antibodies capable of binding to ABP 798/rituximab (Binding Antibody Assay). Samples confirmed to be positive for binding antibodies were subsequently tested in a cell-based assay to determine neutralizing activity against ABP 798/rituximab (Neutralizing Antibody Assay).
  Developing antibody incidence was defined as participants with a negative or no binding antibody result at baseline and a positive antibody result at any post-baseline time point.
Time Frame: Day 1 through the end of study (48 weeks).
Population: Participants with a binding negative or no result at baseline and an available postbaseline result
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 97 | 94 | 97
Participants
  Binding antibody positive | 14 | 13 | 20
  Neutralizing antibody positive | 8 | 4 | 10

24. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Findings
Description: Clinically significant clinical laboratory findings were defined as laboratory results that were ≥ Grade 3, based on the CTCAE version 4.03.
Time Frame: Day 1 through the end of study (48 weeks).
Population: All randomized participants who received at least 1 infusion of study drug (safety analysis set)
Measure: Count of Participants; unit: Participants
Arm/Group | ABP 798 / ABP 798 | Rituximab (EU) / Rituximab (EU) | Rituximab (US) / ABP 798
Number analyzed (Participants) | 104 | 104 | 103
Participants
  Hemoglobin - decrease (anemia) | 0 | 0 | 1
  Lymphocytes - decrease | 64 | 54 | 52
  Alanine aminotransferase - increase | 1 | 0 | 0
  Gamma glutamyl transferase - increase | 5 | 0 | 2
  Potassium - increase (hyperkalemia) | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Dose 1: weeks 1 to 24. Doses 1 and 2: weeks 1 to 48.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Weeks 1-24: ABP 798: Participants received 1000 mg ABP 798 by intravenous infusion on days 1 and 15 (dose 1).
- Weeks 1-24: Rituximab (EU): Participants received 1000 mg rituximab (EU formulation) by intravenous infusion on days 1 and 15 (dose 1).
- Weeks 1-24: Rituximab (US): Participants received 1000 mg rituximab (US formulation) by intravenous infusion on days 1 and 15 (dose 1).
- Weeks 1-48: ABP 798 / ABP 798: Participants received ABP 798 on days 1 and 15 (dose 1) and a second dose of ABP 798 at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
- Weeks 1-48: Rituximab (EU) / Rituximab (EU): Participants received rituximab (EU formulation) on days 1 and 15 (dose 1) and a second dose of rituximab (EU formulation) at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
- Weeks 1-48: Rituximab (US) / ABP 798: Participants received rituximab (US formulation) on days 1 and 15 (dose 1) and transitioned to receive ABP 798 at weeks 24 and 26 (dose 2). Each dose consisted of two 1000 mg intravenous infusions 2 weeks apart.
Arm/Group | Weeks 1-24: ABP 798 | Weeks 1-24: Rituximab (EU) | Weeks 1-24: Rituximab (US) | Weeks 1-48: ABP 798 / ABP 798 | Weeks 1-48: Rituximab (EU) / Rituximab (EU) | Weeks 1-48: Rituximab (US) / ABP 798
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/104 | 0/103 | 0/104 | 0/104 | 0/103
Serious Adverse Events (participants affected / at risk) | 4/104 | 5/104 | 5/103 | 8/104 | 8/104 | 8/103
Other Adverse Events (participants affected / at risk) | 21/104 | 15/104 | 14/103 | 38/104 | 22/104 | 19/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 1-24: ABP 798 (N=104) | Weeks 1-24: Rituximab (EU) (N=104) | Weeks 1-24: Rituximab (US) (N=103) | Weeks 1-48: ABP 798 / ABP 798 (N=104) | Weeks 1-48: Rituximab (EU) / Rituximab (EU) (N=104) | Weeks 1-48: Rituximab (US) / ABP 798 (N=103)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Erythema migrans (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
Sepsis syndrome (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Weeks 1-24: ABP 798 (N=104) | Weeks 1-24: Rituximab (EU) (N=104) | Weeks 1-24: Rituximab (US) (N=103) | Weeks 1-48: ABP 798 / ABP 798 (N=104) | Weeks 1-48: Rituximab (EU) / Rituximab (EU) (N=104) | Weeks 1-48: Rituximab (US) / ABP 798 (N=103)
Nausea (Gastrointestinal disorders) | 4 | 2 | 1 | 8 | 3 | 1
Bronchitis (Infections and infestations) | 3 | 2 | 1 | 7 | 3 | 2
Nasopharyngitis (Infections and infestations) | 5 | 4 | 1 | 9 | 6 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 7 | 8 | 13 | 9 | 11
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 6 | 2 | 3 | 10 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT02792699/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/99/NCT02792699/SAP_001.pdf